CLINICAL TRIAL: NCT02308033
Title: Solubilized Metronidazole And/oR Terconazole Gels Intra-Vaginal Efficacy and Safety
Brief Title: Multi-Center Study of New Medications to Treat Vaginal Infections
Acronym: SMART GIVES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Curatek Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MTC-001 (Trial 2)
Record Dates: First submitted 2014-12-01; First posted 2014-12-04 (Estimated); Results first posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Vaginal Infection
MeSH Terms: conditions — Vaginitis | interventions — Metronidazole; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metronidazole vaginal gel (Active Comparator): One applicator full at bedtime
  Interventions: Drug: Metronidazole
- Gel vehicle (Placebo Comparator): One applicator full at bedtime
  Interventions: Drug: Gel vehicle

INTERVENTIONS:
Drug: Metronidazole
  Arms: Metronidazole vaginal gel
Drug: Gel vehicle
  Arms: Gel vehicle

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of metronidazole gel in the treatment of vaginal infections.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of vaginal infection that is confirmed by laboratory testing and:
* Capable of providing written informed consent or assent
* Currently not menstruating and not anticipating menses during treatment
* If heterosexually active, subject must be post-menopausal for ≥ 1 year, surgically sterile, or practicing an acceptable form of birth control
* Negative pregnancy test
* Other criteria as identified in the protocol

Exclusion Criteria:

* Other infectious causes of vulvovaginitis
* Subject has recently used, or is expected to require the concomitant use of prohibited medications/products
* Nursing mother
* Use of any investigational drug within 30 days of enrollment
* History of hypersensitivity to any ingredient/component of the formulations
* Other criteria as identified in the protocol

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Borgman, Ph.D., Study Director — Curatek Pharmaceuticals
Locations (35):
- United States (35):
  - University of Alabama, Birmingham, Alabama
  - MomDoc Womens Health Research, Scottsdale, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Gossmont Center for Clinical Research, La Mesa, California
  - Genesis Center for Clinical Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Downtown Women's Health Care, Denver, Colorado
  - Red Rocks Ob/Gyn, Lakewood, Colorado
  - Women's Health CT Ob/Gyn, Bridgeport, Connecticut
  - Segal Institute for Clinical Research, North Miami, Florida
  - Discovery Clinical Research, Plantation, Florida
  - Georgia Regents University, Augusta, Georgia
  - Atlanta North Gynecology, Roswell, Georgia
  - Mount Vernon CLinical Research, Sandy Springs, Georgia
  - Rosemark Womens Care Specialists, Idaho Falls, Idaho
  - Women's Health Practice, Champaign, Illinois
  - Women's Healthcare Specialists, PC, Kalamazoo, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Women's Clinic of Lincoln, Lincoln, Nebraska
  - Legacy Women's Health, Las Vegas, Nevada
  - R. Garn Mabey Jr., MD Gynecology, Las Vegas, Nevada
  - Lawrence Ob/Gyn Clinical Research LLC, Lawrenceville, New Jersey
  - Women's Health Research Center, Plainsboro, New Jersey
  - Suffolk OB/GYN, Port Jefferson, New York
  - East Carolina Women's Center, New Bern, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Radiant Research, Columbus, Ohio
  - Drexel University, Philadelphia, Pennsylvania
  - Philapelphia Clinical Research, LLC, Philadelphia, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - James T. Martin, MD, North Charleston, South Carolina
  - The Jackson Clinic, Jackson, Tennessee
  - TMC Life Research, Inc., Houston, Texas
  - Harborview Medical Center, Seattle, Washington
  - Women's Clinical Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Metronidazole Vaginal Gel: One applicator full at bedtime
  Metronidazole
- Gel Vehicle: One applicator full at bedtime
  Gel vehicle
Period: Overall Study
Arm/Group | Metronidazole Vaginal Gel | Gel Vehicle
Started | 102 | 102
Completed | 76 | 83
Not Completed | 26 | 19
Not completed — Normal Gram stain at Baseline | 13 | 10
Not completed — Positive for STD at Baseline | 7 | 4
Not completed — Lost to Follow-up | 6 | 5

BASELINE CHARACTERISTICS:
Population: modified intent-to-treat (mITT) population includes all subjects randomized to treatment and administered at least one dose of study drug. In addition, subjects must have a Nugent score of 4 or more on Baseline visit Gram stain slide.
Groups:
- Total: Total of all reporting groups
Arm/Group | Metronidazole Vaginal Gel | Gel Vehicle | Total
Number analyzed (Participants) | 76 | 83 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (8.76) | 35.8 (10.48) | 34.5 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 83 | 159
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 67 | 74 | 141
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 47 | 45 | 92
  White | 25 | 32 | 57
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 76 | 83 | 159

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure as Assessed by the Investigator at the Test-of-cure Visit
Description: The percentage of participants with clinical cure in each arm was compared. Clinical cure of bacterial vaginosis is defined as 1. discharge has returned to normal/physiologic, 2. the whiff test is negative for any amine "fishy" odor, 3. the saline wet mount is <20% clue cells
Time Frame: 7-14 days after beginning treatment
Population: mITT population (Baseline Gram stain Nugent score of 4 or more and used at least one dose of study medication)
Measure: Count of Participants; unit: Participants
Arm/Group | Metronidazole Vaginal Gel | Gel Vehicle
Number analyzed (Participants) | 76 | 83
Participants | 47 | 18
Statistical Analysis 1: Comparison: Metronidazole Vaginal Gel vs Gel Vehicle; Test type: Superiority; p < 0.001, Chi-squared, Corrected

2. Secondary Outcome: Improvement of BV Clue Cells
Description: Clue cells on wet mount were assessed and categorized as absent (<20%) or present (>=20%). Absence of clue cells is associated with improvement. The comparison was for percentage between arms for clue cells absent (<20%).
Time Frame: 7-14 days after beginning treatment
Population: mITT population (Baseline Gram stain Nugent score of 4 or more and used at least one dose of study medication)
Measure: Count of Participants; unit: Participants
Arm/Group | Metronidazole Vaginal Gel | Gel Vehicle
Number analyzed (Participants) | 76 | 83
Participants
  Clue cells absent | 52 | 19
  Clue cells present | 17 | 58
  Data missing | 7 | 6
Statistical Analysis 1: Comparison: Metronidazole Vaginal Gel vs Gel Vehicle; Test type: Superiority; p < 0.001, Chi-squared, Corrected

3. Secondary Outcome: Microbiologic Improvement/Cure
Description: For bacterial vaginosis (BV), Gram stain Nugent scores are catergized as normal (0 to 3), intermediate (4 to 6) or BV (7 to 10). Normal scores are associated with BV microbiologic cure. The percentage of participants with normal scores were compared between treatments.
Time Frame: 7-14 days after beginning treatment
Population: mITT population (Baseline Gram stain Nugent score of 4 or more and used at least one dose of study medication)
Measure: Count of Participants; unit: Participants
Arm/Group | Metronidazole Vaginal Gel | Gel Vehicle
Number analyzed (Participants) | 76 | 83
Participants
  Normal Nugent score | 38 | 7
  Intermediate Nugent score | 16 | 11
  BV Nugent score | 15 | 59
  Not taken | 7 | 6
Statistical Analysis 1: Comparison: Metronidazole Vaginal Gel vs Gel Vehicle; Comparison of normal Nugent scores at 7-14 days; Test type: Superiority; p < 0.001, Chi-squared, Corrected

4. Secondary Outcome: Number of Participants Reporting Complete Resolution of Symptoms by Test of Cure Visit
Description: Subjects reported if symptoms completely resolved and the date of resolution. The percentage of participants reporting complete resolution of symptoms was compared between arms.
Time Frame: 7-14 days after beginning treatment
Population: mITT population (Baseline Gram stain Nugent score of 4 or more and used at least one dose of study medication)
Measure: Count of Participants; unit: Participants
Arm/Group | Metronidazole Vaginal Gel | Gel Vehicle
Number analyzed (Participants) | 76 | 83
Participants | 43 | 32
Statistical Analysis 1: Comparison: Metronidazole Vaginal Gel vs Gel Vehicle; Comparison of the number of subjects whose reported their symptoms completely resolved; Test type: Superiority; p = 0.034, Chi-squared, Corrected

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Adverse events were collected at study visits, from subject diaries and from spontaneous reports
Time Frame: Any time during study participation (up to 30 days)
Population: The safety population includes all subjects randomized to treatment and administered at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Metronidazole Vaginal Gel | Gel Vehicle
Number analyzed (Participants) | 96 | 97
Participants | 42 | 31

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the entire course of the study (up to 30 days after beginning treatment).
Description: Adverse events were collected through direct questioning at each post-baseline visit, by participant diaries, and by spontaneous reporting. The safety population includes all participants randomized to treatment and administered at least one dose of study drug, and includes subjects who had a normal gram stain Nugent score at the baseline visit.
Arm/Group | Metronidazole Vaginal Gel | Gel Vehicle
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/97
Other Adverse Events (participants affected / at risk) | 25/96 | 10/97
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metronidazole Vaginal Gel (N=96) | Gel Vehicle (N=97)
Vulvovaginal pruritis (Reproductive system and breast disorders) | 8 (8) | 6 (6)
Vulvovaginal candidiasis (Infections and infestations) | 7 (7) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators have the right to disclose and publish results of the Study conducted by them; provided that, in order to protect any Sponsor confidential information, Investigator shall submit to Sponsor manuscripts at least 30 days before submission for publication or 10 days before public presentation. After that time, Investigator is free to submit the manuscript for publication or deliver the presentation, provided Investigator removes any confidential information as directed by Sponsor

DOCUMENTS (2):
  • Study Protocol (2015-03-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT02308033/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT02308033/SAP_001.pdf